CLINICAL TRIAL: NCT06333366
Title: Intra-gastrointestinal Monitoring Device (PDT) to Detect Intra-Abdominal Hypertension (IAH): First-In-Human Study of Feasibility and Safety
Brief Title: First-In-Human Study of PDT to Detect IAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Dotspace Inc. (Industry)
Responsible Party: Principal Investigator, Dong-Ru Ho, Attending Physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202301590A0C501; Application No.2402020052 (Other: Chang Gung Memorial Hospital)
Record Dates: First submitted 2024-02-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Intra-Abdominal Hypertension
Keywords: Intra-Abdominal hypertension; Intravesical pressure; Intra-gastrointestinal monitoring device; laparoscopic surgery; Abdominal compartment Syndrome
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intraabdominal pressure (IAP) monitor (Experimental): Patient who will take laparoscopic surgery will be checked for intra-abdominal pressure, intra-vesical pressure, and intra-gastrointestinal pressure ri-operative stage. PDT passage time will be checked.
  Interventions: Device: Intra-gastrointestinal monitoring device (PDT)

INTERVENTIONS:
Device: Intra-gastrointestinal monitoring device (PDT) — The PressureDOT(PDT) is an active intra-gastrointestinal device, that is intended to be introduced in the gastrointestinal tract, approximately along whole. The device is battery powered. The signal is wirelessly transmitted through outside the body and received by waist receiver, using an antenna array applied to the skin with a protection guard at the level of the abdomen.

SUMMARY:
PDT is a continuous pressure monitoring for Intra-Abdominal hypertension (IAH) designed to be less invasive than pan-endoscopic evaluation, more tolerable than abdominal tapping, and more effective than intravesical pressure measurement for IAH. The PDT device consists of a piezoelectric sensor module with a low power Bluetooth wireless transmitter encased in biocompatible capsule. The device will be swallowed after activation. Following PDT insertion, the patient is fitted with a custom, removable external waist accessory containing a receiver, which is worn during monitoring and provide PDT location by signal analysis with sufficient information to provide IAH trends.

DETAILED DESCRIPTION:
The participant will receive first phantom capsule after complete survey before the test, which include standard clinical intra-vesical pressure measurement in the perioperative period of laparoscopic surgery. The phantom capsule is an equal-weighted device of the same outer shell but without the electric circuits. After the phantom capsule has been passed out, the participant will receive the standard PDT capsule to record measured information continuously. The date of the laparoscopic surgery should be within follow-up day 2 to day 6. Standard clinical intra-vesical pressure measurement will only be applied in the perioperative period of laparoscopic surgery. The participant will still be monitored by standard PDT capsule afterwards. After the PDT capsule passed out, the participant will receive complete checkup again for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patient volunteer planning for laparoscopic surgery
* Subjects willing to sign an informed consent form (ICF),
* Adult subjects, age ≥ 20 and age ≤ 80 years old
* BMI between 15（kg/m2）- 35（kg/m2）
* Subjects willing to comply to study protocol requirements (blood pressure measurement, diet, alcohol, study visits, blood sampling, etc.)
* Patient who had been scheduled for any laparoscopic surgery which may alter intra-abdominal pressure.
* Patient volunteer planning for laparoscopic surgery, as self-declared and confirmed by screening assessments and Principal Investigator's judgment

Exclusion Criteria:

* Patients with a high risk for capsule retention (such as intestinal diverticula, acute abdominal pain without regular defecation indicating intestinal obstruction or a history of abdominal operation or intestinal reconstructed operation),
* Any evidence that occlusion of gastrointestinal tract is obvious or severe paralytic ileus that may result in intra-abdominal hypertension in need of immediate surgical intervention not caused by base of tongue (i.e., central apnea, neurologic disorder, retropalatal collapse, nasal obstruction)
* Any condition that subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Any factor that, in the surgeon's judgment, would pose a risk to surgery or placement of an intra-gastrointestinal monitoring device
* Any factor that, in the surgeon's judgment, would make the subject unlikely to respond to PDT insertion and pressure measurement.
* Congenital anomalies of gastrointestinal tract or any other anatomical abnormality of the head, neck, chest, or abdomen that would be a contraindication to placement of the PDT device and usage of the external device
* There are no exclusion criteria based on gender, race or ethnicity
* Patients with a history of Crohn's disease i* Patients with serious systematic diseases such as congestive heart failure, renal failure or severe liver disease.
* Any blood disorder identified by haematocrit <30% or >55%
* History of hepatitis B, hepatitis C, or HIV
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Female subjects who are pregnant, planning on becoming pregnant or nursing
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Coagulation disorder, wound healing and bleeding disorder or taking anticoagulant medication
* The presence of any other active implanted device, such as cardiac pacemaker or other implanted electro medical devices.
* The presence of any other wireless sensor or transmitter located in abdomen (excluding compatible device also for pressure sensing and other location is acceptable)
* Impaired fasting glucose or impaired glucose tolerance (for Patient volunteer planning for laparoscopic surgery)
* Any contraindication to the use of the PDT system as listed in the device Instructions for Use (IFU) (i.e. any known allergy to PDMS)
* Subject has dysphagia

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-07-16 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of device-related or sensor insertion/removal procedure-related adverse events | 15 days
  evaluating of incidence of adverse event (AE)
Rate of foreign body reaction due intra-gastrointestinal insertion | 15 days
  evaluating GI symptoms
Rate of GI symptoms, i.e. inflammation, infection, diarrhea, bowel obstruction, and ileus | 15 days
  evaluating safety
Incidence of sensor failure | 15 days
  evaluating stability of device

SECONDARY OUTCOMES:
Percentage of users feedback in the form of clinical questionnaire to assess the 'easiness' of insertion procedure with questionnaire | 1 day
  evaluating feed back
Duration of PDT insertion and explantation procedure | 15 days
  monitoring usability needs
Incidence of side effects in Post explantation follow-up | 30 days
  follow up for sequel
Rate of GI dysfunction after 10 days post explantation of the PDT sensor. Follow-up via phone call after 30 days | 30 days
  monitoring of GI symptoms

OTHER OUTCOMES:
Rate of sensor ability to measure intra-gastrointestinal pressure (IGP) to allow the development of the algorithm | 5 days
  workup for correlation
Incidence of influence of interference substances (i.e. water, saliva, gastric juice, bile, intestinal secretion, feces, and food debris ) | 7 days
  evaluating feasibility of working condition

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-Ru Ho, Chiayi City, Taiwan

REFERENCES:
- [Background] Liao CH, Cheng CT, Chen CC, Wang YH, Chiu HT, Peng CC, Jow UM, Lai YL, Chen YC, Ho DR. Systematic Review of Diagnostic Sensors for Intra-Abdominal Pressure Monitoring. Sensors (Basel). 2021 Jul 15;21(14):4824. doi: 10.3390/s21144824. PMID 34300564
- [Result] Liao CH, Cheng CT, Chen CC, Jow UM, Chen CH, Lai YL, Chen YC, Ho DR. An Ingestible Electronics for Continuous and Real-Time Intraabdominal Pressure Monitoring. J Pers Med. 2020 Dec 24;11(1):12. doi: 10.3390/jpm11010012. PMID 33374271